CLINICAL TRIAL: NCT01899092
Title: A Phase I,II Open-Label Dose Escalation Study to Evaluate the Safety and Efficacy of Single Doses of TT-034 for Subjects With Chronic Hepatitis C (CHC) Infection
Brief Title: Safety and Efficacy Study of Single Doses of TT-034 in Patients With Chronic Hepatitis C
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tacere Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2801001
Record Dates: First submitted 2013-07-08; First posted 2013-07-15 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis C
Keywords: Genotype 1; Chronic Hepatitis C; CHC; HCV; Hepatitis; RNAi; shRNA; ddRNAi; AAV8; AAV; Adeno-associated virus; Adeno-associated viral vectors
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic; Hepatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Escalating Dose of TT-034 (Experimental): The study contains one dose escalation arm with active drug.
  Interventions: Drug: TT-034

INTERVENTIONS:
Drug: TT-034 — The study drug will be given as a single dose IV infusion on Day 1. 5 different dose levels corresponding to the 5 cohorts of the study will be given.

SUMMARY:
The study is a first in man, dose escalation study that will measure the safety and efficacy of TT-034 in the treatment of patients with chronic hepatitis C. The study is divided into 5 dose levels. Subjects will be given a single dose delivered by IV infusion. The subjects will be monitored and the data analyzed. After a set time, between 6 and 10 weeks depending on the dose level, the next set of subjects will be dosed. The study drug is a gene therapy treatment that produces molecules that destroy the Hepatitis C virus (HCV) in infected cells. Once the study drug is given, it cannot be withdrawn. Additionally, once an individual receives a dose, he or she will not be able to receive a second dose, but will remain eligible to receive most other HCV treatments.

DETAILED DESCRIPTION:
This is a first-time use of a method of therapy designed to transfer anti-HCV genetic sequences into the hepatocytes of subjects infected with HCV. The anti-HCV sequences will be comprised of three different short hairpin RNAs (shRNA) that have the ability to directly cleave the RNA genome of HCV by a process known as RNA interference. The transfer of the anti-HCV sequences will be accomplished using a "vector" that was made from an adenovirus-associated virus (AAV) by removing the viral genes and replacing them with a non-replicating genetic sequence that produces three different shRNA that target three different regions within the HCV genes. This type of vector has been used in other clinical trials in order to transduce the hepatocytes of subjects who suffer from hemophilia.

ELIGIBILITY:
Inclusion Criteria:

Subjects must a history of chronic HCV infection defined as documented HCV genotype 1 infection for at least 6 months.

* Subjects must have:

  1. Documented failure to respond to prior treatment or relapse with a combination of peg-interferon (peg-IFN), ribavirin (RBV), and either boceprevir or telaprevir, OR a combination of peg-IFN and ribavirin or
  2. Subject is ineligible or unwilling to receive a combination of peg-IFN, RBV, and either boceprevir or telaprevir.
* Female subjects have to be of non-childbearing potential, defined as meeting any of the following criteria:

  1. Female subjects over the age 60.
  2. Female subjects aged 45-60 years old must be amenorrhoeic for at least 2 years and must have serum follicle stimulating hormone (FSH) levels > 30 IU/L.
  3. Female subjects with hysterectomy or bilateral oophorectomy. All female subjects must have a negative serum pregnancy test at Screening and a negative urine pregnancy test at Baseline.
* Male subjects and their partners must be willing to comply with the following requirements to use 2 methods of effective contraception: Male subjects with a vasectomy must use a condom. Without a vasectomy, male subjects must use a condom. The female must be sterile or willing to use an additional form of contraception.
* Baseline HCV RNA level of > 100,000 IU/mL and:
* No evidence of cirrhosis at Screening
* At least 3 months since prior therapy for HCV
* A willingness to enroll in a 5 year follow-up safety study

Exclusion Criteria:

* Body mass index < 18.5 or > 30
* Total body weight > 80 KG
* Female subjects of childbearing potential (including females with tubal ligation) or women who are pregnant or nursing
* Male subjects who are unwilling to provide the required semen samples
* Presence of nAb levels to AAV8 that abrogate AAV8 transduction
* Severe Liver disease
* Hepatocellular carcinoma (HCC) or suspicion of HCC
* Coronary artery disease
* Platelet count of < 150 x 109/L or Creatinine ≥ 1.5 mg/dL at Screening
* Hypertension with systolic blood pressure consistently ≥ 130 mmHg or diastolic blood pressure consistently ≥ 90 mmHg
* Screening examinations indicative of possible occult malignancy unless cancer has been excluded
* Family history of colon cancer in any first-degree relative unless ruled out by colonoscopy
* Positive for human immunodeficiency virus 1 (HIV1) or HIV2 antibody
* Co-infection with hepatitis B virus
* History of autoimmune disease
* Renal impairment
* Hospitalization for liver disease within 60 days of Screening
* Use of drugs of abuse in the prior 3 months
* Other concomitant disease or condition likely to significantly decrease life expectancy or cancer
* Treatment with an investigational drug within 6 months preceding the first dose of trial medication
* Received an AAV vector previously or any other gene transfer agent in the previous 6 months
* History of cardiac abnormalities, as assessed at the Screening Visit
* Twelve-lead ECG demonstrating QTcB > 465 ms at Screening
* Chronic hepatic diseases
* Evidence of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, psychiatric, neurologic, or allergic diseases.
* Evidence of autoimmune disease or pre-existing autoimmune or antibody-mediated diseases
* Use of immunosuppressive medications within 6 months before the entry into this study, except for inhaled or topical corticosteroids

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-01; Primary Completion 2016-09 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
The primary objective is to assess the safety and tolerability of single escalating doses of TT-034 administered IV as a single infusion to subjects with CHC. | 6 months

SECONDARY OUTCOMES:
To assess the activity of TT-034 on the viral load of subjects with CHC receiving single escalating doses of TT-034 | 6 months

OTHER OUTCOMES:
To determine the maximum tolerable dose or the optimal efficacy dose (whichever comes first) | 6 months
To determine the viral load | 6 months
To assess the presence of viral escape mutants in subjects with detectable viral load after receiving TT-034 | 6 months
To monitor TT-034 vector DNA levels and shRNA expression in the target organ (liver) after dosing with TT-034 | 3 weeks
To monitor TT-034 vector DNA levels and shRNA expression peripherally (in blood) after dosing with TT-034 | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David Suhy, PhD, Study Director — Tacere Therapeutics, Inc.
Locations (4):
- United States (4):
  - UCSD Antiviral Research Center, San Diego, California
  - Duke Clinical Research Institute, Durham, North Carolina
  - The Liver Institute at Methodist Dallas, Dallas, Texas
  - The Texas Liver Institute, San Antonio, Texas